CLINICAL TRIAL: NCT06926218
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HSK47388 in Healthy Volunteers
Brief Title: This Study is to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) of HSK47388 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK47388-101
Record Dates: First submitted 2025-03-27; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: HSK47388, Phase I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HSK47388 (Experimental): Single oral doses of HSK47388
  Interventions: Drug: HSK47388
- placebo (Experimental): single oral dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK47388 — cohort 1 to cohort 5
  Arms: HSK47388
Drug: Placebo — cohort 1 to cohort 5
  Arms: placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, SAD study to evaluate the safety, tolerability and PK of HSK47388 in healthy adult participants and preliminarily evaluate the PD of HSK47388

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
2. Adult males and females between ≥ 18 and ≤ 55 years (inclusive) at Screening.
3. Able and willing to attend the necessary visits to the study site

Exclusion Criteria:

1. Participants with any disease history that may affect the safety evaluation or in vivo process of IP as judged by the PI or delegate, including central nervous, cardiovascular, digestive, respiratory, urinary, blood, immune and endocrine diseases. Participants with childhood asthma (resolved) can be included at the discretion of the PI.
2. Underlying physical or psychological medical condition that, in the opinion of the PI or delegate, would make the participant unlikely to comply with the protocol or complete the study per protocol.
3. Participants who may not be able to complete the study for other reasons, cannot comply with the requirements of the study, or are unsuitable to participate in the study as judged by the PI or delegate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | 7 days after single dose
  The incidence, severity, and relationship to IP of AEs. Change from Baseline in clinical laboratory parameters (ie, hematology, serum chemistry, coagulation, and urinalysis parameters), physical examination findings, vital signs

SECONDARY OUTCOMES:
Cmax | Predose up to Day 5 postdose
  Maximum concentration
Tmax | Predose up to Day 5 postdose
  Time to maximum concentration
AUC | Predose up to Day 5 postdose
  Area under the drug concentrationtime curve
t1/2 | Predose up to Day 5 postdose
  Apparent terminal half-life
CL/F | Predose up to Day 5 postdose
  Apparent total plasma clearance of drug

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No